CLINICAL TRIAL: NCT06323486
Title: Effects of Accelerated Bilateral Sequential Theta Burst Stimulation on Dual-task Cost, Depression, Cognition and Other Outcomes in Older Adults With Treatment-resistant Depression: A Randomized, Double-blind, Sham-controlled Trial
Brief Title: Accelerated Bilateral Sequential Theta Burst Stimulation in Older Adults With Treatment-resistant Depression
Acronym: CogniTReaD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Shores Centre for Mental Health Sciences (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-015-B
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Treatment-resistant depression; Accelerated bilateral sequential theta burst stimulation; Repetitive transcranial magnetic stimulation; Motoric-cognitive risk syndrome; Randomized controlled trial; Brain stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: We will enroll patients who are willing to be randomized to either the accelerated bilateral sequential theta burst stimulation (absTBS)-sham or sham-absTBS treatment sequence arms. In the absTBS-sham sequence, participants shall receive the active absTBS treatment at Week 1, followed by sham treatment at Week 3, while in the sham-absTBS sequence, participants shall receive sham treatment at Week 1, followed by the active absTBS treatment at Week 3. The primary rationale for employing this sequential treatment strategy for both arms in this trial is to ensure that those assigned to the sham-absTBS group do not have to wait for longer periods to begin receiving the active absTBS therapy and to maintain blinding continuity.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We shall perform a double-blinding system where the participants, study investigators, transcranial magnetic stimulation (TMS) technicians (those who operate and administer TMS procedures), and research assistants (outcome assessors) are masked to the assignment of the enrolled participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- absTBS-sham treatment sequence arm (Other): Those assigned to the accelerated bilateral sequential theta burst stimulation (absTBS)-sham arm shall receive the blinded active absTBS treatment at Week 1. At Week 3, they shall receive the blinded sham treatment.
  Interventions: Device: active accelerated bilateral sequential theta burst stimulation and sham treatment
- Sham-absTBS treatment sequence arm (Other): In the sham-absTBS arm, the blinded sham treatment shall be administered at Week 1. The blinded active absTBS treatment shall be given at Week 3.
  Interventions: Device: active accelerated bilateral sequential theta burst stimulation and sham treatment

INTERVENTIONS:
Device: active accelerated bilateral sequential theta burst stimulation and sham treatment — We shall use the Magpro device (Magventure) employing the specialized Active/Sham B70 coil.
  absTBS shall be administered consisting of 6 sessions daily (with a 50-minute interval between treatment sessions) on Mondays to Fridays or for a maximum of 5 working days of daily treatment. The target stimulation intensity will be set at 90 to 120% of the subject's resting motor threshold (RMT). Each session shall be composed of administration of continuous theta burst stimulation (triplet burst pulses at 50 Hz, repeated at 5 Hz, for a total of 600 pulses per session over 40 seconds administered on the right dorsolateral prefrontal cortex) and then intermittent theta burst stimulation (triplet burst pulses at 50 Hz bursts, repeated at 5 Hz, 2 s on and 8 s off, for a total of 600 pulses per session over about 3 min, administered on the left dorsolateral prefrontal cortex).
  The sham treatment will be conducted for the same number of sessions and duration as the absTBS treatment sessions.

SUMMARY:
The CogniTReaD study is a pilot clinical trial that will compare the effects of active accelerated bilateral sequential theta burst stimulation (absTBS) and sham or inactive treatment. The goal is to see if absTBS can help older adults with treatment-resistant depression (TRD) by looking at dual-task cost and mood, as well as other cognitive functions, anxiety levels, quality of life, and physical performance, while also checking for any treatment side effects. The study will recruit participants who will receive different study treatments in a specific order. The study will be double-blinded, meaning neither the participants nor the researchers will know who is receiving which treatment. The study will include people who are 50 years old or older and diagnosed with treatment-resistant depression with at least a moderate severity of depression. This study seeks to discover if absTBS can modify a dementia risk marker (i.e., dual-task cost and depression) in older patients with TRD, and to determine the effect size for larger investigations in the future.

DETAILED DESCRIPTION:
The CogniTReaD study is a two-arm, sham-controlled, double-blinded, treatment-sequenced, randomized clinical trial that will evaluate and explore the effects and safety of accelerated bilateral sequential theta burst stimulation (absTBS) compared to sham control in terms of improving dual-task cost, cognitive functions, depression, other outcomes (anxiety, health-related quality of life, activities of daily living, global impression, and other gait performance), and occurrence of adverse events (AE) measured at Week 2 (i.e., posttreatment acute effects) in older adults with treatment-resistant depression (TRD). We shall also evaluate the effects and safety of absTBS on improving dual-task cost, cognitive functions, depression and occurrence of AE in terms of AE occurrences measured at Week 6, Week 8, and Week 10 (i.e., posttreatment delayed effects) in older adults with TRD.

ELIGIBILITY:
Inclusion Criteria

1. Aged 50 years or older;
2. Mini International Neuropsychiatric Interview (MINI)-confirmed diagnosis of a non-psychotic major depressive disorder;
3. Currently in a major depressive episode with a score on HAMD-17 of 17 or more;
4. Insufficient response (i.e., failure to achieve remission) to at least two appropriate courses of antidepressant medications during the current depressive episode (i.e., meeting the criteria for TRD);
5. Participants taking or not taking any psychotropic medication/s. If the eligible participant is on any psychotropic medications, the participant should have taken the medication/s at a stable dose for at least 1 week before the start of study intervention treatment and be willing to remain on a stable dose throughout the study follow-up;
6. Passing the TMS safety screen; and
7. Those who have the capacity to provide consent and who voluntary consent to participate in the study.

Exclusion Criteria

1. Those with MINI-confirmed active substance use disorder within the last 3 months;
2. Those with lifetime MINI-confirmed diagnosis of bipolar I disorder, delusional disorder, schizophrenia, schizoaffective disorder, or schizophreniform disorder;
3. Those with major unstable medical comorbidities (i.e., rapidly deteriorating medical/neurological conditions that poses a significant risk to a person's life);
4. Those with a diagnosis of dementia confirmed using the Global Clinical Dementia Rating (CDR) with a score greater than or equal to 1.
5. Those with significant neurological conditions, such as those with any disease process associated with increased intracranial pressure, space-occupying intracranial lesion, history of epilepsy/seizure except those induced by ECT, or febrile seizure of infancy or a single occurrence of seizure associated with a known drug, cerebral aneurysm, or major head trauma resulting to loss of consciousness more than 5 minutes;
6. Those with cardiac pacemaker or implanted mediation pump;
7. Those with intracranial implants/hardwares, including but not limited to aneurysm clips, shunts, stimulators, cochlear implants, electrodes, or any other metal material inside or near the head (excluding the mouth) that cannot be safely removed;
8. Those who are taking more than 2 mg of Lorazepam daily (or equivalent) or taking any dose of an anticonvulsant that may potentially hamper rTMS efficacy;
9. Those who are unable to express and understand using the English language; and
10. Individuals who are pregnant or who are likely pregnant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Dual-task Cost | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Hamilton Depression Rating Scale 17 (HAMD-17) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Adverse events (AE) | Week 1, Week 2, Week 3, Week 6, Week 8, and Week 10
  An AE is defined as any untoward medical occurrence associated with any of the study interventions (active absTBS or sham) whether or not considered related to the study intervention.
  A serious AE to any serious and unforeseen occurrence related or possibly related to the participation in the study that can lead to hospitalization, disability, or death.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-Cognitive-13 (ADAS-Cog-13) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Alzheimer's Disease Assessment Scale-Cognitive-13 (ADAS-Cog-13) plus modalities score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Trail Making A (TMT-A) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Trail Making B (TMT-B) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Digit Symbol Substitution Test (DSST) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Digit Span Forward (DSF) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Digit Span Backward (DSB) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Category Verbal Fluency (CVF) score | Week 0 (baseline), Week 2, Week 6, Week 8, and Week 10
Change in Montreal Cognitive Assessment (MoCA) score | Week 0 (baseline), Week 2
Change in Colour Word Interference Test (CWIT) score | Week 0 (baseline), Week 2
Change in Patient Health Questionnaire-9 (PHQ-9) score | Week 0 (baseline), Week 2
Change in Geriatric Depression Scale 30 (GDS-30) score | Week 0 (baseline), Week 2
Change in Generalized Anxiety Disorder 7 (GAD-7) score | Week 0 (baseline), Week 2
Change in Short Form 36 (SF-36) score | Week 0 (baseline), Week 2
Change in Alzheimer Disease Cooperative Study - Activities of Daily Living inventory (ADCS-ADL) score | Week 0 (baseline), Week 2
Change in Lawton-Brody Instrumental Activities of Daily Living (LB-IADL) score | Week 0 (baseline), Week 2
Change in Clinical Global Impression (CGI) score | Week 0 (baseline), Week 2
Change in Short Physical Performance Battery (SPPB) score | Week 0 (baseline), Week 2
Change in Timed Up & Go (TUG) score | Week 0 (baseline), Week 2

CONTACTS AND LOCATIONS:
Overall Officials: Amer M. Burhan, MBChB, MSc, Principal Investigator — Ontario Shores Centre for Mental Health Sciences and University of Toronto
Locations (1):
- Ontario Shores Centre for Mental Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data can be made available by request from qualified researchers/investigators.